CLINICAL TRIAL: NCT02840331
Title: Pilot Study on Intra-abdominal Photodynamic Diagnosis in Peritoneal Carcinosis
Acronym: Hypericin-PDT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Beckert, Chief consultant, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hypericin-PDT
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Peritoneal Carcinomatosis
Keywords: Gastric carcinoma; Peritoneal carcinomatosis; Photodynamic diagnosis; Photodynamic therapy; St. John's Wort; Peritoneal metastasis
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms | interventions — Hypericum extract LI 160; LAIF 900; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- St. John's Wort & PDD, PDT (Experimental): St. John's Wort 900 milligram once oral preoperative & intraoperative irradiation with light (photodynamic diagnosis (PDD) and therapy (PDT), with the appropriate wavelength (390-440 nanometer) over 15 minutes
  Interventions: Drug: St. John's Wort; Device: Photodynamic diagnostic and therapy

INTERVENTIONS:
Drug: St. John's Wort — Single oral doses (900 milligram) 2-4 hours before laparoscopy
  Other Names: Laif 900
Device: Photodynamic diagnostic and therapy — Intraoperative irradiation with light (photodynamic diagnosis (PDD) and therapy (PDT), with the appropriate wavelength (390-440 nanometer) over 15 minutes

SUMMARY:
The study would examine by hypericin-supported Fluoreszenzlaparoskopy in terms of tumor size, number and location of the combination of photodynamic diagnosis (PDD) and therapy (PDT) with regard to the detection of peritoneal metastases of locally advanced gastric cancer at 50 adult patients.

DETAILED DESCRIPTION:
Hypericin-PDT study is an examination of patients with gastric cancer. The peritoneal carcinosis (PC) of the adult represents the final stage of an advanced tumor and was treated in the past, usually by means of palliative chemotherapy. An improvement in survival for patients with PC could be further improved through the use of maximum cytoreductive surgery (CRS) can be achieved with radical removal of the entire tumor mass and the combination of CRS and intraperitoneal hyperthermic chemotherapy (HIPEC) event-free survival and overall survival. A cure of patients is achieved only in the rarest cases. An essential problem in the treatment of peritoneal carcinomatosis is that can only be poorly differentiated from surrounding tissue due to their location, the tumors often not well recognized because of their size or. This results to differ (as scar tissue) for the surgeon the difficulty between eigentlichem tumor tissue and surrounding tissue.

Through the use of innovative diagnostic and therapeutic options (for example, photodynamic diagnosis (PDD) and therapy (PDT)) above mentioned problems can be improved. In photodynamic diagnosis contrast between tumor and surrounding healthy tissue is improved by an interaction of photodynamic active substance with light of a particular wavelength. The PDT is based on a topical or systemic administration of a photosensitizer (here hypericin), which is irradiated with light of a suitable wavelength and in the presence of oxygen oxygen radicals (with the consequence of a direct cytotoxicity of the tumor cells leading) forms.

The study will be carried out in the Department of General, Visceral and Transplantation Surgery Tübingen at 50 adult patients. The study proposed would examine by hypericin-supported Fluoreszenzlaparoskopy in terms of tumor size, number and location of the combination of photodynamic diagnosis (PDD) and therapy (PDT) with regard to the detection of peritoneal metastases of locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Computertomography - morphologically locally - advanced gastric cancer (Classification of Malignant Tumours (TNM): size or direct extent of the primary tumor > 3 or degree of spread to regional lymph nodes positive) without distant metastases (except peritoneum)
* Histologically confirmed adenocarcinoma of the stomach
* Karnofsky Index > 70

Exclusion Criteria:

* Patients who are considered inoperable because of a reduced general condition:

  * Congestive heart failure (New York Heart Association (NYHA) Functional Classification III / IV),
  * Severe coronary heart disease, non-treatable arrhythmia or non-adjustable hypertension,
  * Severe asthma suffering (Chronic obstructive pulmonary disease)
* Distant metastases except peritoneum
* Patients with a contraindication related to the present study
* Allergy or intolerance to the study drug or a substance with chemical similarity to the study medication.
* Lack of capacity to consent
* Participation in another interventional therapy studies at intervals of 30 days
* Contraindication to taking the prescribed study medication the physician's discretion
* Pregnancy/ Breastfeeding
* Women in childbearing age who refuse:

  * Simultaneously apply two appropriate contraceptive measures or maintain a full hetero-sexual abstinence at least 28 days prior to the study and for at least 28 days after administration of study medication
  * To stop breast-feeding during the study and through 6 months after the end of study
* Men who refuse:

  - To use a latex condom during any sexual contact with childbearing women during the study and at least 28 days after completion of study, even if they are successful vasectomy.
* - Sperm donor to make up at least 28 days after completion of study.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Peritoneal metastases in terms of tumor size [centimeter, cm] | Day 1 (day of surgery)
  Detection of peritoneal metastases of locally - advanced gastric cancer by hypericin - supported Fluoreszenzlaparoskopie in terms of tumor size [cm]
Peritoneal metastases in terms of number [n] | Day 1 (day of surgery)
  Detection of peritoneal metastases of locally - advanced gastric cancer by hypericin - supported Fluoreszenzlaparoskopie in terms of number [n]
Peritoneal metastases in terms of location | Day 1 (day of surgery)
  Detection of peritoneal metastases of locally - advanced gastric cancer by hypericin - supported Fluoreszenzlaparoskopie in terms of location [central, right upper, epigastrium, left upper, , left flank, left lower, pelvis, riht lower, right flank, upper jejunum, lower jejunum, upper ileum, lower illeum]

SECONDARY OUTCOMES:
Hypericin level | Day 1 (day of surgery)
  Hypericin levels in the peritoneum and serum the day of surgery
Histological evidence of apoptosis | Day 1 (day of surgery)
  Histological evidence of apoptosis in peritoneal metastasis after photodynamic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Beckert, Prof. Dr., Principal Investigator — University Department of General, Visceral and Transplant Surgery
Locations (1):
- University Department of General, Visceral and Transplant Surgery, Tübingen, Baden.Württemberg, Germany

IPD SHARING:
Plan to Share IPD: No